CLINICAL TRIAL: NCT00544466
Title: Allogeneic Stem Cell Transplant With a Novel Conditioning Therapy Using Helical Tomotherapy, Melphalan, and Fludarabine in Hematological Malignancies
Brief Title: Helical Tomotherapy, Fludarabine Phosphate, and Melphalan Followed By Allo-HSCT in Hematological Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04199; P30CA033572 (NIH); CHNMC-04199; CDR0000570241 (Registry Identifier: NCI PDQ); NCI-2010-00355 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: acute myeloid leukemia with multilineage dysplasia following myelodysplastic syndrome; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; recurrent adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary acute myeloid leukemia; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine phosphate; Melphalan; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzyme inhibitor, radiation therapy, transplant) (Experimental): PREPARATIVE REGIMEN*: Patients receive fludarabine phosphate IV on days -7 to -3 and melphalan IV on day -2. Patients also undergo helical tomotherapy twice daily on days -7 to -4. TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0. NOTE: *Treatment begins 2 days earlier in patients receive tacrolimus and/or sirolimus for GVHD prophylaxis.
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: fludarabine phosphate — 25 mg/m2 day -7 through day -3 prior to transplant
Drug: melphalan — 140 mg/m2 day -2 prior to transplant
Procedure: allogeneic hematopoietic stem cell transplantation — Cells infused on Day 0 of transplant regimen
Radiation: intensity-modulated radiation therapy — Each fraction is 150 cGy, 2 fractions each day on day -7 through day -4 prior to transplant

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as fludarabine phosphate and melphalan, and HT before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving HT together with fludarabine phosphate and melphalan before a transplant may stop this from happening.

PURPOSE: This clinical trial studies helical tomotherapy (HT), fludarabine phosphate, and melphalan followed by donor stem cell transplant in treating patients with hematologic malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess the feasibility in terms of toxicity and safety of HT in combination with Fludarabine (fludarabine phosphate) and Melphalan as a preparative regimen for allogeneic stem cell transplantation in patients with Hematological Malignancies: acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), and myelodysplastic syndromes (MDS).

SECONDARY OBJECTIVES: I. To evaluate within the confines of this pilot study, incidence of neutrophil and platelet engraftment, survival on day +180, the overall survival, and disease free survival in patients with Hematological Malignancies: ALL, AML, and MDS.

II. To evaluate incidence of primary and secondary engraftment failure, incidence of relapse, incidence of acute and chronic transplant related complications, including veno-occlusive disease of the liver (VOD), organ toxicity, secondary malignancies, including treatment-related myelodysplastic syndrome, and acute and chronic graft-versus-host disease (GVHD), as well as post-transplant chimerism.

OUTLINE: PREPARATIVE REGIMEN*: Patients receive fludarabine phosphate intravenously (IV) on days -7 to -3 and melphalan IV on day -2. Patients also undergo HT twice daily on days -7 to -4.

TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0. NOTE: *Treatment begins 2 days earlier in patients receive tacrolimus and/or sirolimus for GVHD prophylaxis.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Recipient, or recipient's parents, or recipient's legal guardians must have signed a voluntary, informed consent in accordance with institutional and federal guidelines
* Must have histopathologically confirmed diagnosis in one of the followed categories:

  * AML
  * MDS with intermediate or high-risk disease
  * ALL
* Children and adults at any age with significant morbidity, as determined by the primary bone marrow transplant (BMT) doctor (MD), and approved by the principal investigator (PI)
* Able to lie supine in a full body cast for approximately 30 minutes, the anticipated duration of each treatment session; for younger patients deep conscious sedation may be required
* Performance status evaluated by Zubrod or Karnofsky (KPS) Performance Scales in patients > 16 years or Lanksy Performance Scale in children =< 16 years must have a score >= 70%
* Adequate cardiac function: cardiac ejection fraction > 50% by multi gated acquisition scan (MUGA) scan and/or by echocardiogram
* Adequate pulmonary function: adults (older than 16 years): diffusing capacity of carbon monoxide (DLCO) > 50%; for young children in whom pulmonary function tests (PFT) are not applicable: assessment by a pediatrician or pulmonary consult
* Adequate renal function as demonstrated by: creatinine clearance or glomerular filtration rate (GFR) > 60 cc/min (24 hour urine collection)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) =< 5.0 times the institutional upper limits of normal
* Patients must have less than 15% peripheral blasts
* Pre-treatment tests must have been preformed within 30 days prior to initiation of high-dose chemotherapy
* No other medical and/or psychosocial problems, which in the opinion of the primary physician or principle investigator would place the patient at unacceptable risk from this regimen

Exclusion Criteria:

* Patients with Acute Undifferentiated Leukemia (AUL), i.e. no lymphoid or myeloid markers
* Previous radiation therapy to more than 20% of bone marrow containing areas, or to any area exceeding 2000 cGy
* Patients with Fanconi Anemia
* Major medical or psychiatric disorders that would seriously compromise patient tolerance of this regimen
* Human immunodeficiency virus (HIV) infection
* Evidence of Hepatitis B or C infection or evidence of cirrhosis
* Uncontrolled viral, bacterial or fungal infection
* Patients with recent (within 4 weeks) serious viral, fungal, or bacterial infection are excluded
* Patients with radiographic changes indicating pulmonary disease, including but not limited to: pulmonary nodules, infiltrates, pleural effusion are excluded unless cleared by pulmonary biopsy showing no evidence for active pulmonary disease

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-07-31 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2025-12-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rosenthal, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 75 patients, who consented to the study, 13 of them became ineligible after screening. So only 62 patients received the study treatment.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant)
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients consented to the study.
Arm/Group | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant)
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 55 [9 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 62
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 and Above Toxicities of Helical Tomotherapy (HT) in Combination With Fludarabine and Melphalan Followed by Allogeneic Stem Cell Transplantation.
Description: Toxicities (adverse events) were evaluated using the modified Bearman Scale and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 100 days post treatment
Measure: Number; unit: events
Arm/Group | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant)
Number analyzed (Participants) | 62
events | 793

2. Secondary Outcome: Overall Survival on Day 180 Days Post-transplant
Description: Overall survival (OS) was measured from peripheral stem cell infusion to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula. Participants were followed up to 180 days after transplant and Kaplan-Meier survival analysis was used to generate the Overall Survival estimate at 180 days.
Time Frame: Up to 180 days post-transplant
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant)
Number analyzed (Participants) | 62
Percent Probability | 81 [68 to 89]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to Day 100 post-transplant. All-Cause Mortality was assessed from start of protocol treatment to death due to any cause, or last follow-up, whichever comes first, assessed up to 12 years.
Arm/Group | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant)
All-Cause Mortality (participants affected / at risk) | 43/62
Serious Adverse Events (participants affected / at risk) | 13/62
Other Adverse Events (participants affected / at risk) | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant) (N=62)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (2)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 1 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (4)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 5 (7)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 1 (1)
Fistula, GI (Gastrointestinal disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 7 (7)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (2)
Infection, Bacterial (Infections and infestations) | 1 (1)
Infection, Fungal (Infections and infestations) | 1 (1)
Infection, Viral (Infections and infestations) | 2 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 3 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (3)
Calcium, serum-low (hypocalcemia) (Investigations) | 1 (1)
Creatinine (Investigations) | 4 (4)
Glucose, serum-high (hyperglycemia) (Investigations) | 3 (3)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 3 (3)
Potassium, serum-low (hypokalemia) (Investigations) | 2 (2)
Proteinuria (Investigations) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 2 (2)
Apnea (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Intra-operative injury (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Radiation Therapy, Transplant) (N=62)
Coagulation - Other (Specify, __) (Blood and lymphatic system disorders) | 3 (4)
Edema:head and neck (Blood and lymphatic system disorders) | 14 (14)
Edema:limb (Blood and lymphatic system disorders) | 29 (30)
Edema:trunk/genital (Blood and lymphatic system disorders) | 3 (3)
Edema:viscera (Blood and lymphatic system disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 19 (23)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI (Blood and lymphatic system disorders) | 11 (14)
Hemorrhage, GU (Blood and lymphatic system disorders) | 16 (17)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 16 (17)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 3 (3)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Blood and lymphatic system disorders) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 19 (24)
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 14 (14)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20 (20)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 13 (13)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 7 (7)
Platelets (Blood and lymphatic system disorders) | 20 (26)
Portal vein flow (Blood and lymphatic system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 4 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 4 (4)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 3 (3)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 2 (2)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 34 (35)
Hypotension (Cardiac disorders) | 18 (20)
Left ventricular diastolic dysfunction (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 6 (6)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 18 (22)
Valvular heart disease (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Neuroendocrine: gonadotropin secretion abnormality (Endocrine disorders) | 1 (1)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 2 (2)
Parathyroid function, low (hypoparathyroidism) (Endocrine disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Nystagmus (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 43 (45)
Ascites (non-malignant) (Gastrointestinal disorders) | 8 (8)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 56 (57)
Distension/bloating, abdominal (Gastrointestinal disorders) | 13 (13)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 10 (10)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 13 (13)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 10 (10)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 13 (13)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 18 (18)
Hemorrhoids (Gastrointestinal disorders) | 6 (6)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 5 (5)
Incontinence, anal (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 42 (45)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 34 (48)
Nausea (Gastrointestinal disorders) | 60 (61)
Necrosis, GI (Gastrointestinal disorders) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 2 (2)
Perforation, GI (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 7 (7)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1)
Ulcer, GI (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 46 (47)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 45 (46)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (4)
Hypothermia (General disorders) | 1 (1)
Insomnia (General disorders) | 17 (17)
Pain (General disorders) | 58 (216)
Pain - Other (Specify, __) (General disorders) | 6 (14)
Rigors/chills (General disorders) | 15 (15)
Sweating (diaphoresis) (General disorders) | 1 (1)
Weight gain (General disorders) | 24 (24)
Weight loss (General disorders) | 12 (12)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 2 (2)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
Allergy/Immunology - Other (Specify, __) (Immune system disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 9 (10)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 11 (11)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 24 (42)
Infection - Other (Specify, __) (Infections and infestations) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 8 (16)
Infection with unknown ANC (Infections and infestations) | 4 (6)
Infection, Bacterial (Infections and infestations) | 25 (41)
Infection, Fungal (Infections and infestations) | 8 (8)
Infection, Viral (Infections and infestations) | 13 (14)
Viral hepatitis (Infections and infestations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 49 (52)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 50 (52)
Acidosis (metabolic or respiratory) (Investigations) | 6 (6)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 58 (62)
Alkaline phosphatase (Investigations) | 37 (39)
Alkalosis (metabolic or respiratory) (Investigations) | 9 (9)
Amylase (Investigations) | 1 (1)
Bicarbonate, serum-low (Investigations) | 8 (8)
Bilirubin (hyperbilirubinemia) (Investigations) | 13 (13)
CPK (creatine phosphokinase) (Investigations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Investigations) | 19 (19)
Calcium, serum-low (hypocalcemia) (Investigations) | 56 (60)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 23 (23)
Creatinine (Investigations) | 29 (29)
Glucose, serum-high (hyperglycemia) (Investigations) | 53 (54)
Glucose, serum-low (hypoglycemia) (Investigations) | 9 (9)
Magnesium, serum-high (hypermagnesemia) (Investigations) | 20 (20)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 59 (59)
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 17 (17)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 46 (47)
Potassium, serum-high (hyperkalemia) (Investigations) | 19 (19)
Potassium, serum-low (hypokalemia) (Investigations) | 54 (57)
Proteinuria (Investigations) | 10 (11)
Sodium, serum-high (hypernatremia) (Investigations) | 8 (8)
Sodium, serum-low (hyponatremia) (Investigations) | 57 (57)
Syndromes - Other (Specify, __) (Investigations) | 3 (3)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 51 (53)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 9 (9)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 4 (4)
Confusion (Nervous system disorders) | 20 (21)
Dizziness (Nervous system disorders) | 10 (11)
Encephalopathy (Nervous system disorders) | 1 (1)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Mental status (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 37 (52)
Neurology - Other (Specify, __) (Nervous system disorders) | 3 (3)
Neuropathy: cranial (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 4 (4)
Neuropathy: sensory (Nervous system disorders) | 13 (14)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 8 (8)
Seizure (Nervous system disorders) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 17 (17)
Bladder spasms (Renal and urinary disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 3 (3)
Incontinence, urinary (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 5 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 11 (11)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Flushing (Skin and subcutaneous tissue disorders) | 4 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 15 (15)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 18 (18)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 39 (40)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 43 (45)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 5 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes